CLINICAL TRIAL: NCT06672978
Title: A Multi-Center, Open-Label, Single-Arm, Phase 2 Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Vabomere (Meropenem-Vaborbactam) In The Treatment Of Children With Complicated Urinary Tract Infection, Including Acute Pyelonephritis
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Meropenem-Vaborbactam in Children With Complicated Urinary Tract Infection, Including Acute Pyelonephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rempex (a wholly owned subsidiary of Melinta Therapeutics, LLC) (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: Melinta Therapeutics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML-VAB-201-3248-2; 2024-516360-29 (EudraCT Number); U1111-1310-7249 (Other: Universal Trial Number)
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Acute Pyelonephritis; Complicated Urinary Tract Infection
MeSH Terms: interventions — meropenem and vaborbactam; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Age 6 to < 12 years (Experimental): Participants will receive meropenem-vaborbactam via an IV infusion for a minimum of 3 days, for up to 14 days.
  Participants with clinical improvement have the option to switch to an oral antibiotic or home IV therapy after Day 3.
  Interventions: Drug: Meropenem-Vaborbactam; Drug: Antibiotics
- Cohort 2: Age 2 to < 6 years (Experimental): Participants will receive meropenem-vaborbactam IV infusion for a minimum of 3 days, for up to 14 days.
  Participants with clinical improvement have the option to switch to an oral antibiotic or home IV therapy after Day 3.
  Interventions: Drug: Meropenem-Vaborbactam; Drug: Antibiotics
- Cohort 3: Age 3 months to < 2 years (Experimental): Participants will receive meropenem-vaborbactam IV infusion for a minimum of 3 days, for up to 14 days.
  Participants with clinical improvement have the option to switch to an oral antibiotic or home IV therapy after Day 3.
  Interventions: Drug: Meropenem-Vaborbactam; Drug: Antibiotics

INTERVENTIONS:
Drug: Meropenem-Vaborbactam — Administered as specified in the treatment arm
  Other Names: Vabomere
Drug: Antibiotics — Administered as prescribed by the study physician in accordance with local guidelines and regulations.

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of meropenem-vaborbactam administered by intravenous (IV) infusion in children 3 months and above to less than 12 years with complicated urinary tract infections (cUTI), including acute pyelonephritis (AP).

ELIGIBILITY:
Key Inclusion Criteria:

* Have a clinically suspected and/or bacteriologically documented cUTI or AP judged by the Investigator to require hospitalization for treatment with at least 3 days of IV antibiotics.
* Evidence of pyuria, confirmed by either of the following:

  * A urine specimen that is positive for leukocyte esterase via urine dipstick or urinalysis, or
  * A urine specimen with either > 10 white blood cells (WBCs) per microliter from an unspun urine or > 5 WBCs per high power field from a centrifuged specimen
* Symptomatic or asymptomatic cUTI or AP as specified in the protocol.
* Acute Pyelonephritis (qualifying symptoms specified in protocol).
* Have a pretreatment "baseline" urine specimen obtained for culture by an acceptable method, including suprapubic aspiration (SPA), clean urethral catheterization, in dwelling urethral catheter, or mid-stream clean catch (urine specimens obtained from externally placed urine bags will not be allowed) within 48 hours before the start of the administration of the first dose of IV study drug therapy.
* Must, based on the judgment of the Investigator, require hospitalization initially and 7 to14 days of antibacterial therapy for the treatment of the presumed cUTI.

Key Exclusion Criteria:

* History of hypersensitivity or allergic reaction to beta-lactam antibiotics (for example [e.g.], cephalosporins, penicillins, carbapenems, monobactams).
* Known Vabomere-resistant gram-negative organism from study-qualifying urine or blood culture, confirmed cUTI or AP only due to gram-positive organism from study-qualifying urine or blood culture, or known or suspected infection with organisms that are not adequately covered by Vabomere (e.g., viral, mycobacterial, fungal).
* Receipt of a potentially effective antibacterial drug therapy for cUTI for a duration of more than 24 hours during the previous 72 hours prior to enrollment. Exceptions: participants with unequivocal clinical evidence of treatment failure (that is, worsening signs and symptoms); urine culture confirms resistance to the initial antibiotic; or the participant developed signs and symptoms of cUTI or AP while on antibiotics for another indication.
* Participants undergoing dialysis or with estimated glomerular filtration rate (eGFR) < 30 mL/minute/1.73 m^2, as calculated using the updated bedside Schwartz formula.
* Evidence of significant hepatic disease or dysfunction, including known acute viral or inactive chronic hepatitis or hepatic encephalopathy, or aspartate aminotransferase or alanine aminotransferase > 3 × upper limit normal (ULN), or total bilirubin > 1.5 × ULN.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 28 days

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Day 1 and Day 3: Up to 3 hours post-dose
Time to Maximum Observed Plasma Concentration (Tmax) | Day 1 and Day 3: Up to 3 hours post-dose
Area Under the Plasma Concentration Curve from Zero to Infinity (AUC0-inf) | Day 1 and Day 3: Up to 3 hours post-dose
Overall Response (OR) | Up to 14 days
  OR as assessed by the combined per-participant clinical cure and favorable microbiological response.
Clinical Cure | Up to 14 days
  Clinical cure is defined as the complete resolution or significant improvement of signs and symptoms of cUTI or AP present at baseline, no new symptoms, and participant is alive.
Favorable Microbiological Response (Microbiological Eradication) | Up to 14 days
  Favorable microbial response is defined as the reduction of baseline pathogen(s) (< 10^3 colony-forming units per milliliter [CFU/mL] and at least 1-log reduction from baseline) or negative urine culture, negative repeated blood culture if blood culture was positive for pathogen(s) growth at baseline, and participant is alive.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Melinta Therapeutics, LLC
Locations (24):
- United States (4):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - University of Nebraska Medical Center, Department of Pediatrics, Omaha, Nebraska
  - University Hospitals Rainbow Babies & Children's Hospital, Cleveland, Ohio
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment "Sv. Ivan Rilski - 2003" OOD, Department of Pediatric Diseases, Dupnitsa
  - Multiprofile Hospital for Active Treatment "Dr. Tota Venkova", Gabrovo, Department of Pediatrics Diseases, Gabrovo
  - Multiprofile Hospital for Active Treatment - Pazardzhik, Second Department of Pediatric Diseases, Pazardzhik
  - University Multipurpose Hospital for Active Treatment "Sveti Georgi", Pediatrics Clinic, Plovdiv
  - University Multiprofile Hospital for Active Treatment 'Kanev', Ruse, Department of Pediatrics, Rousse
  - Multiprofile Hospital for Active Treatment "Dr. Ivan Seliminski", Sliven, Sliven
  - Multiprofile Hospital For Active Treatment, "Vita", Department of Urology, Sofia
  - University Hospital for Active Treatment and Emergency Medicine (UHATEM) "N. I. Pirogov" LTD, Urology Clinic, Department of Urology, Sofia
- University Hospital for Infectious Diseases "Dr. Fran Mihaljevic", Zagreb, Croatia
- Georgia (6):
  - JSC Vian, Batumi
  - Geo Hospitals LLC, Tbilisi
  - JSC Georgian Clinics, Tbilisi
  - LTD L. Managadze National Center of Urology, Tbilisi
  - New Hospitals LLC, Tbilisi
  - Vian JSC, Tbilisi
- Greece (3):
  - University Hospital Alexandroupolis, Department of Pediatrics, Alexandroupoli
  - Agia Sofia Children's Hospital, Infectious Diseases, Pediatrics - General, Athens
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Poland (2):
  - St. Jadwiga the Queen Provincial Hospital #2 in Rzeszow, 1st Teaching Department of Pediatrics and Pediatric Gastroenterology, Pediatric Cardiology Subdivision, Rzeszów
  - St. Hedwig of Silesia Hospital in Trzebnica, Pediatric Department with Infantible Sub-department, Trzebnica

IPD SHARING:
Plan to Share IPD: No